CLINICAL TRIAL: NCT00910728
Title: A PhaseI/II, Open Label Multi-Centre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the JAK2 Inhibitor AZD1480 Administered Orally to Patients With Primary Myelofibrosis (PMF) and Post-Polycythaemia Vera/Essential Thrombocythaemia Myelofibrosis (Post-PV/ET MF
Brief Title: Study to Assess the Safety of AZD1480 in Patients With Myeloproliferative Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: University of Texas (Other); New York City Hoffman Center (Unknown); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D1060C00001
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Primary Myelofibrosis (PMF); Post-Polycythaemia Vera; Essential Thrombocythaemia Myelofibrosis
Keywords: Primary Myelofibrosis (PMF); Post-Polycythaemia Vera/Essential Thrombocythaemia Myelofibrosis (Post-PV/ET MF); Myeloproliferative diseases; Phase I; Phase II; Bone marrow
MeSH Terms: conditions — Primary Myelofibrosis | interventions — AZD 1480

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD1480
  Interventions: Drug: AZD1480

INTERVENTIONS:
Drug: AZD1480 — Oral capsule 2.5 mg, 10 mg and 40 mg

SUMMARY:
This study is being conducted to test study drug AZD1480 to see how it may work to treat myeloproliferative diseases. The main purpose of this study is to determine the safety and tolerability of AZD1480. This is the first time the drug has been given to humans and is classed as a first time in man study. Its main purpose is to establish a safe dosage of the drug and provide additional information on any potential side effects this drug may cause. The study will also assess the blood levels and action of AZD1480 in the body over a period of time and will indicate whether the drug has a therapeutic effect on myeloproliferative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myelofibrosis requiring therapy
* Evidence of post-menopausal status or sterile
* ECOG Performance Status </=2

Exclusion Criteria:

* Prior therapy with any JAK2 medications
* Significant lung disorder or lung disease
* Previous radiation therapy to chest wall or chest infection requiring antibiotic treatment within 28 days before study screening
* Eye disease of the cornea
* Patients requiring oxygen supplementation
* Ejection fraction <45% (ECHO/MUGA) or significant pulmonary hypertension >40 mm Hg (by Echo/Doppler)
* Forced Expiratory Volume (FEV1)/Forced Vital Capacity (FVC) <70% predicted or >130% predicted
* Diffusing capacity of the Lung for Carbon Monoxide (DLCO) corrected for hemoglobin <60% predicted, oxygen saturation <88% at rest or after a 6-minute flat walk, without supplemental oxygen
* Chest infection requiring antibiotics within 7 days of the first dose of Investigational product.

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-05; Primary Completion 2012-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — MDACC; Ronald Hoffman, MD, Principal Investigator — Mt. Sinai; Vincent Ribrag, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Becker Hewes, MD, Study Director — AstraZeneca
Locations (3):
- United States (2):
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Research Site, Villejuif, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Commenced 19MAY2009. All subjects recruited to Part A only (based on emerging data). 65 patients were enrolled of which 35 recieved at least 1 dose of AZD1480.
Pre-assignment Details: Patients ≥25 years of age with primary myelofibrosis (MF) and post-polycythaemia vera/essential thrombocythaemia MF who had relapsed, were intolerant of, or were refractory to MF-directed therapy were enrolled.
Groups:
- 2.5 mg QD; 5.0 mg QD; 10 mg QD; 30 mg QD; 50 mg QD; 70 mg QD; 10 mg BID; 15 mg BID; 20 mg QD: AZD1480 may be administered orally in capsules
Period: Overall Study
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 50 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 20 mg QD
Started | 6 | 3 | 3 | 3 | 6 | 1 | 6 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not Completed | 6 | 3 | 3 | 3 | 5 | 1 | 6 | 3 | 3
Not completed — Lack of Efficacy | 2 | 3 | 1 | 2 | 1 | 0 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0
Not completed — (not specified) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 70 mg QD | 15 mg BID | 30 mg QD | 50 mg QD | 10 mg BID | 20 mg QD | Total
Number analyzed (Participants) | 6 | 3 | 3 | 1 | 4 | 3 | 6 | 6 | 3 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (7.7) | 66.3 (9.6) | 76.7 (10.5) | 56.0 (0) | 66.5 (10.3) | 49.3 (4.2) | 69.3 (3.8) | 65.3 (11.3) | 75.7 (3.8) | 65.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 0 | 1 | 5 | 2 | 2 | 14
  Male | 5 | 2 | 2 | 0 | 4 | 2 | 1 | 4 | 1 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters Following Single Dosing: AUC0-12
Description: Single dose AUC0-12 (ug*h/L)
Time Frame: 0 to 12 hour sampling (Day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post dose)
Population: Pharmacokinetic.
  Note - no GeoCV(%) was captured in the TFL. Hence the geometric mean was still presented as applicable but with the SD (since only available).
Measure: Geometric Mean (Standard Deviation); unit: ug*h/L
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 6 | 4 | 6 | 3
ug*h/L | 69.2 (27.5) | 295 (68.2) | 278 (257) | 1860 (546) | 5800 (0) | 425 (190) | 497 (191) | 3090 (2060) | 472 (257)

2. Primary Outcome: Pharmacokinetic Parameters Following Single Dosing: AUC0-24
Description: Single dose AUC0-24 (ug*h/L)
Time Frame: 0 to 24 hour sampling (Day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose)
Population: Pharmacokinetic.
  Note - no GeoCV(%) was captured in the TFL. Hence the geometric mean was still presented as applicable but with the SD (since only available).
  From the BID schedule we can not derive the single dosing AUC0_24 and hence this is not presented/calculated.
Measure: Geometric Mean (Standard Deviation); unit: ug*h/L
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 0 | 0 | 6 | 3
ug*h/L | 70.2 (28.7) | 308 (76) | 285 (252) | 2000 (624) | 6260 (0) |  |  | 3540 (2570) | 508 (280)

3. Primary Outcome: Pharmacokinetic Parameters Following Single Dosing:AUC0-inf
Description: Single dose AUC(0 to infinity) (ug*h/L)
Time Frame: 0 to 24 hour sampling (Day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose)
Population: Pharmacokinetic.
  Note - no GeoCV(%) was captured in the TFL. Hence the geometric mean was still presented as applicable but with the SD (since only available).
  From the BID (twice a day dosing schedules) we can not derive the PK parameter AUC0_inf following single dosing. With that these do not contribute.
Measure: Geometric Mean (Standard Deviation); unit: ug*h/L
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 0 | 0 | 6 | 3
ug*h/L | 83.5 (36.6) | 312 (79.5) | 378 (290) | 2040 (657) | 6300 (0) |  |  | 3650 (2980) | 517 (294)

4. Primary Outcome: Pharmacokinetic Parameters Following Multiple Dosing: Cmax,ss
Description: Multiple dose Cmax,ss (ug/L)
Time Frame: On Days 1 and 28 at 0, 0,5, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose, and at 0, 2, 4 hours post dose on Days 4 and 10
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ug/L
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 1 | 5 | 4 | 5 | 3
ug/L | 51.3 (18) | 134 (36.3) | 176 (179) | 658 (265) | 1500 (0) | 218 (72.3) | 334 (68.2) | 924 (461) | 241 (346)

5. Primary Outcome: Pharmacokinetic Parameters Following Multiple Dosing: Cmin,ss
Description: Multiple dose Cmin,ss (ug/L)
Time Frame: On Days 1 and 28 at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose and at 0, 2, 4 hours post-dose on Days 4 and 10.
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ug/L
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 6 | 4 | 6 | 3
ug/L | 69.2 (27.5) | 295 (68.2) | 278 (257) | 1860 (546) | 5800 (0) | 425 (190) | 497 (191) | 3090 (2060) | 472 (257)

6. Primary Outcome: Pharmacokinetic Parameters Following Single Dosing: Cmax
Description: Single dose Cmax (ug/L)
Time Frame: 0 to 24 hour sampling (Day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ug/L
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 6 | 4 | 6 | 3
ug/L | 69.9 (32.7) | 133 (54.7) | 157 (145) | 739 (307) | 2600 (0) | 273 (62.2) | 324 (79.5) | 1320 (379) | 268 (227)

7. Primary Outcome: Pharmacokinetic Parameters Following Single Dosing: Vz/F
Description: Single dose Vz/F (L)
Time Frame: 0 to 24 hour sampling (Day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose)
Population: Pharmacokinetic.
  Note - no GeoCV(%) was captured in the TFL. Hence the geometric mean was still presented as applicable but with the SD (since only available).
  Due to the nature of the dosing schedule this PK parameter was not reported for the BID (twice daily dosing) groups.
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 0 | 0 | 6 | 3
L | 222 (125) | 108 (28.1) | 138 (161) | 97 (15) | 57.9 (0) |  |  | 105 (82.2) | 284 (92.3)

8. Primary Outcome: Pharmacokinetic Parameters Following Single Dosing: CL/F
Description: Single dose CL/F (L/h)
Time Frame: 0 to 24 hour sampling (Day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 6 | 4 | 6 | 3
L/h | 35.2 (13.9) | 16 (4.25) | 34.8 (22.5) | 14.7 (5.52) | 11.1 (0) | 22.6 (9.05) | 29.7 (13) | 13.8 (8.5) | 38.7 (16.7)

9. Primary Outcome: Pharmacokinetic Parameters Following Multiple Dosing: CLss/F
Description: Multiple dose CLss/F (L/h)
Time Frame: On Days 1 and 28 at 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours post dose and at 0, 2, 4 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 1 | 5 | 4 | 6 | 3
L/h | 37.8 (6) | 15.8 (4.4) | 30.1 (21.7) | 17 (5.26) | 9.57 (0) | 20 (6.91) | 20.4 (13.8) | 16 (8.94) | 20.8 (21)

10. Primary Outcome: Pharamcokinetic Parameters Following Single Dosing: Tmax
Description: Single dose Tmax (h)
Time Frame: 0 to 24 hour sampling (Day 1: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose)
Measure: Median (Full Range); unit: h
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 6 | 4 | 6 | 3
h | 0.625 [0.5 to 1.5] | 0.75 [0.5 to 2] | 0.75 [0.5 to 0.75] | 1 [1 to 1.5] | 0.75 [0.75 to 0.75] | 0.625 [0.5 to 1] | 0.875 [0.5 to 1] | 0.89 [0.75 to 1.5] | 0.75 [0.5 to 1.03]

11. Primary Outcome: Pharamcokinetic Parameters Following Multiple Dosing: Tmax,ss
Description: Multiple dose Tmax,ss (h)
Time Frame: On Days 1 and 28 at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose and at 0, 2, 4 hours post-dose on Days 4 and 10
Measure: Median (Full Range); unit: h
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 6 | 4 | 6 | 3
h | 0.5 [0.5 to 1] | 0.78 [0.75 to 1] | 0.77 [0.75 to 1] | 0.75 [0.52 to 1] | 1.5 [1.5 to 1.5] | 1 [0.5 to 1.5] | 0.875 [0.75 to 1.5] | 0.78 [0.25 to 2.25] | 1 [0.75 to 3]

12. Primary Outcome: Inhibition of PSTAT3 (Count)
Description: PSTAT3 inhinition
Time Frame: 2hrs and 4 hrs post dose
Measure: Number; unit: # patients with 50% reduction in PSTAT3
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 30 mg QD | 70 mg QD | 10 mg BID | 15 mg BID | 50 mg QD | 20 mg QD
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 1 | 6 | 4 | 6 | 3
# patients with 50% reduction in PSTAT3
  2 Hours post dose | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
  4 Hours post dose | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout study continuously and 30 days post discontinuation of treatment
Arm/Group | 2.5 mg QD | 5.0 mg QD | 10 mg QD | 70 mg QD | 15 mg BID | 20 mg QD | 30 mg QD | 50 mg QD | 10 mg BID
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/3 | 0/3 | 0/1 | 1/4 | 3/3 | 0/3 | 4/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 1/1 | 4/4 | 3/3 | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg QD (N=6) | 5.0 mg QD (N=3) | 10 mg QD (N=3) | 70 mg QD (N=1) | 15 mg BID (N=4) | 20 mg QD (N=3) | 30 mg QD (N=3) | 50 mg QD (N=6) | 10 mg BID (N=6)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ATRIAL FLUTTER/FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 2.5 mg QD (N=6) | 5.0 mg QD (N=3) | 10 mg QD (N=3) | 70 mg QD (N=1) | 15 mg BID (N=4) | 20 mg QD (N=3) | 30 mg QD (N=3) | 50 mg QD (N=6) | 10 mg BID (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
NEUTROPENIUA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
WEIGHT INCREASE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1/1 (1) | 1/1 (1) | 0/0 (0) | 1/1 (1) | 1/1 (1) | 1/1 (1) | 1/1 (1) | 2/2 (2)
PYREXIA (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTHERMIA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OEMEMA PERIPHERAL (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA AGGRAVATED (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATARAC (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
KERATITI (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECCHYMOSI (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC MURMUR (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PARAESTHES (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
EPITAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other